CLINICAL TRIAL: NCT05455606
Title: A Cluster Randomized Trial Comparing an Educationally Enhanced Genomic Tumor Board (EGTB) Intervention to Usual Practice to Increase Evidence-Based Genome-Informed Therapy
Brief Title: Does the Use of a Genomic Tumor Board Increase the Number of Patients Who Receive Genome-Informed Treatment
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: S2108CD; NCI-2022-04626 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); S2108CD (Other: SWOG); SWOG-S2108CD (Other: DCP); S2108CD (Other: CTEP); UG1CA189974 (NIH)
Record Dates: First submitted 2022-07-06; First posted 2022-07-13 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Advanced Malignant Solid Neoplasm; Metastatic Malignant Solid Neoplasm; Recurrent Malignant Solid Neoplasm; Refractory Malignant Solid Neoplasm
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Practice Guidelines as Topic; Standard of Care; Early Intervention, Educational; Educational Status; Methods; Genetic Profile; Interviews as Topic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (usual care) (Active Comparator): Participants receive usual care. This consists of physicians ordering GTT for patients and reviewing the results without the GTB being involved.
  Interventions: Other: Best Practice; Other: Chart Abstraction; Procedure: Genomic Profile; Other: Interview; Other: Questionnaire Administration
- Arm 2 (EGTB) (Experimental): Patients and physicians receive the EGTB intervention. This is comprised of 2 components: the structured GTB and the supporting education. Physicians submit cases for discussion to the GTB within 2 weeks of GTT results. The GTB sessions are held weekly and conducted virtually over a video-conferencing platform. Each case presentation is 10 to 15 minutes long, and 4 to 6 cases are discussed during each 60 minute GTB session. GTT results and clinical data are presented and expert interpretation of genomic test results is provided to help prioritize potential treatment options and provide a framework for interpretation. Supporting education materials are also available online to participants to support GTT decision making.
  Interventions: Other: Chart Abstraction; Other: Educational Intervention; Procedure: Genomic Profile; Other: Interview; Other: Questionnaire Administration; Other: Tumor Board Review

INTERVENTIONS:
Other: Best Practice — Receive usual care
  Other Names: standard of care; standard therapy
  Arms: Arm 1 (usual care)
Other: Chart Abstraction — Ancillary studies
Other: Educational Intervention — Physicians access genomic testing education materials
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
  Arms: Arm 2 (EGTB)
Procedure: Genomic Profile — Patients undergo genomic testing
  Other Names: genetic profile; Genome Profile; Genomic Profiling; Genomic Test; Genomic Testing
Other: Interview — Ancillary studies
Other: Questionnaire Administration — Ancillary studies
Other: Tumor Board Review — Patients undergo genomic tumor board review
  Other Names: multidisciplinary opinion
  Arms: Arm 2 (EGTB)

SUMMARY:
This clinical trial studies how well an educationally enhanced genomic tumor board (EGTB) intervention works to increase the number of patients with solid tumors that have come back (recurrent), do not respond to treatment (refractory), have spread to other parts of the body (metastatic), or are newly diagnosed and spread to other parts of the body (advanced) who receive genome-informed treatment. Genome-informed treatment refers to treatment based on the information found in genomic tumor test results. This study compares the usual approach to reviewing genomic tumor test results with the approach of having a genomic tumor board (GTB) review the test results. A GTB is team of doctors and scientists that have experience in understanding genomic changes and review genomic tumor test results. The tumor board helps to suggest whether there are other cancer treatment options based on patient genetic test results. The usual approach is to review genomic tumor test results without the GTB being involved. This study may help researchers learn if using a GTB enhances the treatment decision making process within 6 months of joining the study. This study may also help researchers learn if using the GTB increases doctors' understanding of genomic tumor test results and increases doctors' comfort level with genomic tumor tests.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine whether an EGTB intervention compared to usual practice increases the proportion of patients who receive evidence-based genome-informed therapy within 6 months after registration to the study.

SECONDARY OBJECTIVES:

I. To compare physician genomic confidence and physician experience with genomic tumor testing (GTT) between arms at baseline and end of study.

II. To compare clinical outcomes between arms by assessing patient survival and time to treatment discontinuation.

III. To compare physician assessment of evidence-based genome-informed therapy to the central study team determination of evidence-based genome-informed therapy, both overall and separately by arm.

IMPLEMENTATION OBJECTIVES:

I. To assess the utilization of GTT and implementation of the EGTB intervention into clinic workflow in order to better understand barriers and facilitators at Recruitment Centers assigned to the active intervention arm using a mixed-methods approach.

II. To assess the evolution of GTT utilization within clinic workflows at recruitment centers assigned to the usual practice (control) arm using a mixed-methods approach.

OUTLINE: Study clinics are randomized to 1 of 2 arms. Participants receive interventions based on this randomization.

ARM 1: Participants receive usual care. This consists of physicians ordering GTT for patients and reviewing the results without the GTB being involved.

ARM 2: Patients and physicians receive the EGTB intervention. This is comprised of 2 components: the structured GTB and the supporting education. Physicians submit cases for discussion to the GTB within 2 weeks of GTT results. The GTB sessions are held weekly and conducted virtually over a video-conferencing platform. Each case presentation is 10 to 15 minutes long, and 4 to 6 cases are discussed during each 60 minute GTB session. GTT results and clinical data are presented and expert interpretation of genomic test results is provided to help prioritize potential treatment options and provide a framework for interpretation. Supporting education materials are also available online to participants to support GTT decision making.

Physicians are followed until the end of the study or through 6 months after their last patient was registered to the study, whichever is later. Patients are followed for 24 months after registration or until a criterion for removal from protocol participation is met, whichever comes first.

ELIGIBILITY:
Inclusion Criteria:

* RECRUITMENT CENTERS INCLUSION
* A Recruitment Center is defined as an outpatient clinic, or group of clinics, belonging to the same National Cancer Institute Community Oncology Research Program (NCORP) or minority/underserved (MU)-NCORP, who will be contributing physicians and patient participants to the study
* Recruitment Centers must be part of an NCORP or MU-NCORP site with Cancer Care Delivery Research (CCDR) funding as this study is supported by CCDR funding. Each clinic included in the Recruitment Center must be associated with Cancer Therapy Evaluation Program (CTEP) site identification (ID).
* Recruitment Centers must send large panel next generation sequencing genomic tests on at least 10 unique patients per month.
* Recruitment Centers must have at least 4 practicing oncologists (including medical, gynecologic, or neuro-oncologists) at the site willing to participate in the study and register within three months of study activation.
* Recruitment Centers must be willing to register a total of 66 patients (over 2 years) to the study.
* Centers must be able to send at least one member of the study team to attend the Recruitment Center's cases presented to the S2108CD Genomic Tumor Board, should the Recruitment Center be randomized to the intervention arm.
* Recruitment Centers must be willing and able to document the number of unique patients on which GTT is ordered at the Recruitment Center and submit this monthly to the S2108CD Study Team.
* PHYSICIAN PARTICIPANT INCLUSION
* Physician participant must be a registering investigator of the Recruitment Center that is participating in the study. If the physician is a registering investigator at more than one Recruitment Center, he/she must choose one Recruitment Center to identify with and enroll patients from.
* Physician participants must be board-eligible or board-certified in Medical Oncology, Gynecologic Oncology, or Neurology with certification or eligible for certification in Neuro-oncology.
* Physician participants must be willing to offer participation in the study to all eligible patients under their care for the duration of the study. A single physician may enroll multiple patients on the study.
* Physician participants must be willing to complete all study questionnaires and, as part of the implementation objective, participate in interviews if invited.
* Physician participants must complete all baseline questionnaires prior to registration.
* Physician participants at a Recruitment Center randomized to the intervention arm must be willing to participate in the educationally enhanced GTB (EGTB).
* PATIENT PARTICIPANT INCLUSION
* Patient participants must have either recurrent, relapsed, refractory, metastatic, or newly diagnosed advanced stage III or stage IV solid tumor malignancy.
* Patient participants must be under the care of a physician enrolled on the study.
* Patient participants may have started anti-cancer treatment for the current diagnosis. The treating physician anticipates that the patient will start a new anti-cancer treatment (either first or subsequent lines) within 6 months after registration.
* Patient participants are allowed to be co-enrolled on other clinical trials including non-treatment studies and studies that include investigational drugs. Patients may be enrolled on genome-informed therapeutic trials, such as LungMAP, MATCH, TAPUR, etc.
* Patient participants' genomic tumor test must have been ordered within 7 days prior to registration with results pending. The genomic testing may be a commercially available panel (such as FoundationOne, Caris, Tempus, etc.) or a non-commercial tumor panel performed at an academic medical center.

  * NOTE: Qualifying GTTs are defined as Clinical Laboratory Improvement Act (CLIA)-certified next generation sequencing (NGS) tissue or liquid biopsy panels, including hotspot, whole gene, deoxyribonucleic acid (DNA) and ribonucleic acid (RNA) (including expression data) panels. Fluorescence-in-situ hybridization (FISH) and immunohistochemistry test results assessing cancer-relevant proteins (e.g. Her2/neu, ALK, MET) and immune parameters (e.g. PD-L1 tests) are also permissible if performed in the context of a larger panel that includes NGS or expression profiling. These tests can come from any commercial or academic laboratory within the United States (US) and they should be ordered with the intent to influence genome-informed treatment decision. Oncotype DX and other panels used for making treatment decisions based on a prognostic read-out (e.g. liquid biopsy minimal residual disease [MRD]) are not permitted.
* Patient participants must be at least 18 years of age.
* Patient participants must have a Zubrod performance status of 0-2.
* Participants (patients and physicians) must sign and give written informed consent in accordance with institutional and federal guidelines. For patient participants with impaired decision-making capabilities, legally authorized representative may sign and give informed consent on behalf of study participants in accordance with applicable federal, local, and Central Institutional Review Board (CIRB) regulations. Documentation of informed consent via remote consent is permissible.

Exclusion Criteria:

* RECRUITMENT CENTERS EXCLUSION
* Recruitment Centers must not have or utilize an existing Genomic Tumor Board (GTB). For the purposes of this study, a Genomic Tumor Board is defined as an interdisciplinary team of clinicians and scientists that reviews genomic testing results and provides guidance on treatment options based primarily on genomic data to the treating physician. The existence of a general multidisciplinary tumor board that addresses all aspects of patient care and treatment is not considered an exclusion criterion. A general multidisciplinary tumor board is defined as an interdisciplinary team of clinicians that primarily discusses all aspects of cancer care, including diagnostic aspects (pathology and radiology), therapeutic options (surgical, radiation and medical) as well as palliative and psychosocial support options.
* PATIENT PARTICIPANT EXCLUSION
* Patient participants must not be going on hospice care at the time of registration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1284 (Actual)
Dates: Start 2022-10-14 (Actual); Primary Completion 2026-12-15 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Percent of patients who receive a treatment that targets a genomic variant for which there is sufficient data to support actionability | Within 6 months of study completion
  Evidence-based genome-informed therapy is defined as the use of a treatment that targets a genomic variant for which there is sufficient data to support actionability. This is a patient-specific measure determined through blinded central review of patient data, following the schemas in the protocol. An independent panel of investigators blinded to the study arm assignment of the study participant will evaluate redacted data from each subject for determination of the primary endpoint. Data supporting the primary endpoint are obtained from the genomic tumor test results PDF, pathology report, primary tumor type, and the S2108CD Treatment Form as well as curated evidence plus evidence level (tier) designation from the Jackson Labs Clinical Knowledge Base.

SECONDARY OUTCOMES:
Physician genomic confidence | Baseline and month 27 after study activation
  Measured by 3-item scale assessing physician confidence in genomic knowledge and ability to explain genomic concepts/make treatment recommendations. This assessment is on the S2108CD Genomic Testing Questionnaire.
Physician experience using genomic tumor testing (GTT) in practice | Baseline and month 27 after study activation
  The physician experience using genomic tumor testing in practice will be assessed using selected items from the National Survey of Precision Medicine in Cancer Treatment, included on the S2108CD Genomic Testing Questionnaire.
Overall survival | From registration until death due to any cause, assessed up to 24 months
  Overall survival on study will be measured from registration until death due to any cause.
Overall survival on new anticancer therapy | From the time new anticancer therapy is initiated on study until deathdue to any cause, assessed up to 24 months
  Overall survival on new anticancer therapy will be measured from the time new anticancer therapy is initiated on study until death due to any cause.
Time to treatment discontinuation | From registration until the last dose recorded or death, assessed up to 24 months
  Time to treatment discontinuation on study will be measured as the time from registration until the last dose recorded or death.
Time to treatment discontinuation on new anticancer therapy | From registration until the last dose recorded or death, assessed up to 24 months
  time to treatment discontinuation on new anticancer therapy will be measured as the time from registration until the last dose recorded or death.

CONTACTS AND LOCATIONS:
Overall Officials: Jens Rueter, Principal Investigator — SWOG Cancer Research Network
Locations (72):
- United States (70):
  - Cancer Center at Saint Joseph's, Phoenix, Arizona
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Hawaii Cancer Care - Westridge, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - HaysMed University of Kansas Health System, Hays, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Olathe Health Cancer Center, Olathe, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - University of Kansas Health System Saint Francis Campus, Topeka, Kansas
  - Saint Joseph Hospital East, Lexington, Kentucky
  - Saint Joseph London, London, Kentucky
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Saint Joseph Mercy Brighton, Brighton, Michigan
  - Saint Joseph Mercy Chelsea, Chelsea, Michigan
  - Ascension Saint John Hospital, Detroit, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Minnesota Oncology - Burnsville, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Fairview Lakes Medical Center, Wyoming, Minnesota
  - Parkland Health Center - Farmington, Farmington, Missouri
  - Truman Medical Centers, Kansas City, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - University of Kansas Cancer Center at North Kansas City Hospital, North Kansas City, Missouri
  - Delbert Day Cancer Institute at PCRMC, Rolla, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - Missouri Baptist Outpatient Center-Sunset Hills, Sunset Hills, Missouri
  - FirstHealth of the Carolinas-Moore Regional Hospital, Pinehurst, North Carolina
  - Essentia Health Cancer Center-South University Clinic, Fargo, North Dakota
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Saint Joseph's/Candler - Bluffton Campus, Bluffton, South Carolina
  - Gibbs Cancer Center-Gaffney, Gaffney, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - MGC Hematology Oncology-Union, Union, South Carolina
  - Ascension Southeast Wisconsin Hospital - Elmbrook Campus, Brookfield, Wisconsin
  - Ascension Saint Francis - Reiman Cancer Center, Franklin, Wisconsin
  - Ascension Columbia Saint Mary's Hospital Ozaukee, Mequon, Wisconsin
  - Ascension Medical Group Southeast Wisconsin - Mayfair Road, Wauwatosa, Wisconsin
- Puerto Rico (2):
  - Doctors Cancer Center, Manatí
  - Centro Comprensivo de Cancer de UPR, San Juan